CLINICAL TRIAL: NCT00456859
Title: Carbonaceous Oral Adsorbent's Effects on Progression of Chronic Kidney Disease (CAP-KD)
Brief Title: Carbonaceous Oral Adsorbent's Effects on Progression of Chronic Kidney Disease
Acronym: CAP-KD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute for Health Outcomes and Process Evaluation Reseach (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAP-KD ver.3
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2007-10-18 (Estimated); Status verified 2007-10

CONDITIONS: Kidney Failure, Chronic
Keywords: chronic kidney disease; oral carbonaceous adsorbent; randomized clinical trial; composite endpoint
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — AST 120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Kremezin

SUMMARY:
The CAP-KD trial is a prospective, multicenter, randomized, open-label, two-arm, parallel group comparison clinical trial and will be conducted as a researcher-directed study to assess the efficacy of Kremezin in preventing the progression of CKD. We compare two groups of patients: those receiving conventional treatment alone and those receiving such treatment paired with Kremezin.

DETAILED DESCRIPTION:
A clinical trial to evaluate the efficacy of the oral carbonaceous adsorbent Kremezin in preventing the progression of chronic kidney disease (the Carbonaceous Oral Adsorbent's Effects on Progression of Chronic Kidney Disease [CAP-KD] trial) in predialysis patients. In the trial we are comparing two treatments: conventional treatment comprising an ACEI and/or ARB together with a low-protein diet, and combination treatment comprising the conventional treatment paired with Kremezin. Furthermore, we will compare the QOL in both groups of patients

ELIGIBILITY:
Inclusion Criteria:

* The subject is an outpatient.
* The subject is 20 years of age or older at the time of consent to participate in the study.
* The subject's serum creatinine value is 5.0 mg/dl or less at the time of case registration.
* The inverse serum creatinine value, calculated using measurements at four or more time points during an observation period that occurs within 48 weeks of case registration, is decreasing, on average, according to linear-regression analysis performed at the case registration center.
* The subject's blood pressure is well controlled before the initial serum creatinine measurement during the observation period.
* The subject has been treated with an ACEI and/or ARB before the initial serum creatinine measurement during the observation period.
* The subject has undergone low-protein diet therapy (> 0.8 g/kg per day) before the initial serum creatinine measurement during the observation period.
* The subject has not changed the type or dose of medication for renal failure for 4 weeks prior to case registration.
* The subject has participated in thorough consultation and has been informed as to the purpose, description, expected adverse effects, and risks of this study according to the consent form, and has voluntarily signed the informed consent form.

Exclusion Criteria:

* The subject has a passage disorder of the gastrointestinal tract.
* The subject has been treated with Kremezin within the period from the initial measurement of the serum creatinine level prior to case registration to the time of study commencement.
* The subject has rapid progressive glomerular nephritis, hydronephrosis, occlusive urinary tract injury, drug-induced nephropathy, or transplanted kidney.
* The subject has complications such as severe hepatopathy, liver cirrhosis, severe infection, class III or above New York Heart Association (NYHA) congestive heart failure, severe arrhythmia, or unstable angina.
* The subject has had cardiac infarction, cerebral infarction, or cerebral hemorrhage within the past 6 months.
* The subject presents with severe nephrotic syndrome (serum albumin < 2 g/dl).
* The subject is currently pregnant, or plans to become pregnant during the study period.
* The subject abuses alcohol.
* The subject has a body weight less than 80% or more than 160% of the standard weight {[height(m)]^2 x 22}.
* The subject has significant difficulty in controlling his/her blood sugar level within 3 months of case registration (hemoglobin [Hb]A1c > 8.0% on one occasion).
* The subject has a progressive malignant tumor.
* The subject is not available for study visits at least once per 2 months to provide urine samples.
* The subject is inappropriate for participation in the study for other reasons, as determined by an investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2004-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The composite primary endpoint comprises the following events:
Doubling of serum Creatinine
Increase in serum Creatinine to 6.0 mg/dl or more
Endstage renal disease (ESRD; defined as that requiring dialysis or renal transplantation)
Death

SECONDARY OUTCOMES:
Variation in urinary protein
Changes in Creatinine Clearance
Changes in health-related quality of life (HRQOL)
Occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yasushi Asano, Study Chair — Jichi Medical University
Locations (1):
- iHope International, Tokyo, Japan

REFERENCES:
- [Background] Morita S, Fukuhara S, Akizawa T, Asano Y, Kurokawa K. Study design and methods for a clinical trial of an oral carbonaceous adsorbent used to prevent the progression of chronic kidney disease (CAP-KD). Clin Exp Nephrol. 2005 Sep;9(3):219-27. doi: 10.1007/s10157-005-0358-7. PMID 16189630
- [Derived] Akizawa T, Asano Y, Morita S, Wakita T, Onishi Y, Fukuhara S, Gejyo F, Matsuo S, Yorioka N, Kurokawa K; CAP-KD Study Group. Effect of a carbonaceous oral adsorbent on the progression of CKD: a multicenter, randomized, controlled trial. Am J Kidney Dis. 2009 Sep;54(3):459-67. doi: 10.1053/j.ajkd.2009.05.011. Epub 2009 Jul 17. PMID 19615804